CLINICAL TRIAL: NCT06264674
Title: A 12-week Double-blind, Multicentre, Randomised, Active-controlled, 2-arm, Parallel-group Clinical Trial to Evaluate the Safety of CHF5993 pMDI 200/6/12.5 μg HFA-152a, Compared to CHF5993 pMDI 200/6/12.5 μg HFA-134a, in Subjects With Asthma.
Brief Title: Comparison Between CHF5993 pMDI 200/6/12.5 µg HFA-152a VS CHF5993 pMDI 200/6/12.5 µg HFA-134a in Subjects With Asthma (TRECOS).
Acronym: TRECOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-05993AB6-03; 2023-503333-22-00 (Other: EMA CTIS); 17142179 (Other: ISRCTN)
Record Dates: First submitted 2023-11-13; First posted 2024-02-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Double-blind multicentre, randomised, active-controlled, 2-arm, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind multicentre, randomised, active-controlled, 2-arm, parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaler CHF5993 200/6/12.5 μg pMDI HFA-152a (Experimental): Active ingredients: BDP/FF/GB 200/6/12.5 μg per actuation; Excipients: HFA-152a propellant.
  Interventions: Drug: CHF5993 200/6/12.5 μg pMDI HFA-152a
- Inhaler CHF5993 200/6/12.5 μg pMDI HFA-134a (Active Comparator): Active ingredients: BDP/FF/GB 200/6/12.5 μg per actuation; Excipients: HFA-134a propellant.
  Interventions: Drug: Inhaler CHF5993 200/6/12.5 μg pMDI HFA-134a

INTERVENTIONS:
Drug: CHF5993 200/6/12.5 μg pMDI HFA-152a — Pressurised Metered Dose Inhaler-2 inhalations twice daily
  Other Names: HFA-152a propellant
  Arms: Inhaler CHF5993 200/6/12.5 μg pMDI HFA-152a
Drug: Inhaler CHF5993 200/6/12.5 μg pMDI HFA-134a — Pressurised Metered Dose Inhaler-2 inhalations twice daily
  Other Names: HFA-134a propellant
  Arms: Inhaler CHF5993 200/6/12.5 μg pMDI HFA-134a

SUMMARY:
The CLI-05993AB6-03 Study is an interventional study designed to investigate the safety and efficacy of a new low global warming potential propellant (HFA-152a) compared to the currently approved one (HFA-134a) in the medication (CHF5993) in patients with moderate to severe asthma

DETAILED DESCRIPTION:
Outpatients attending the hospital clinics/study centers will be recruited. Moderate to severe controlled asthma adult subjects will be recruited. A total of 513 subjects will be randomised. The whole study will last approximately 16 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study related procedure;
* Male and female adults aged ≥ 18 and ≤ 75;
* Body mass index (BMI) within the range of 18.0 to 35.0 kg/m2 inclusive;
* Non-smokers or ex-smokers who smoked < 10 pack-years (pack-years = the number of cigarette packs per day x the number of years) and stopped smoking > 1 year (6 months for e-cigarettes) prior to screening;
* Diagnosis of asthma: physician-diagnosed asthma for at least
* 6 months and with diagnosis before the age of 50 years;
* Stable asthma therapy: a stable treatment with medium/high doses of inhaled corticosteroids (ICS) + long-acting β-agonist (LABA) + long-acting muscarinic antagonist (LAMA) (fixed or free combination) or medium/high doses of ICS+LABA (fixed or free combination) for at least 4 weeks before screening (medium and high-dose ICS defined as BDP non-extrafine > 500-1000 μg and > 1000 μg respectively, or estimated clinical comparable dose).
* Subjects must have a cooperative attitude and the ability to be trained to use correctly the pMDI inhalers and e-Diary, to be able to read/write, to be able to perform the required outcomes measurements (e.g., technically acceptable spirometry, e-Diary completion) and the ability to understand the risks involved.

Exclusion Criteria:

* History of near fatal asthma, hospitalisation for asthma in intensive care unit which in the judgement of the Investigator may place the subject at undue risk, emergency room access for asthma in the previous 6 months before enrolment;
* Asthma exacerbation requiring systemic corticosteroids (SCS) or emergency room admission or hospitalisation within 4 weeks prior to study entry and/or during the run-in period (to be checked again prior to randomisation);
* Non-permanent asthma: exercise-induced, seasonal asthma (as the only asthma-related diagnosis) not requiring daily asthma control medecine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 836 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Relative change from pre-dose Forced Expiratory Volume in one second with (FEV1) (Safety Assessment to evaluate of the potential bronchoconstriction of the study treatment) | Day 1
  Relative change from pre-dose in FEV1 at the 10 min post-dose timepoint

SECONDARY OUTCOMES:
To complete the evaluation of FEV1 and the potential for bronchoconstriction of the study treatment (relative change from pre-dose FEV1) | Day 1, Day 7, Week 4, Week 12
  Relative change from pre-dose in FEV1 at all the post dose timepoints
To complete the evaluation of FEV1 and the potential for bronchoconstriction of the study treatment (absolute change from pre-dose FEV1) | Day 1, Day 7, Week 4, Week 12
  Absolute change from pre-dose in FEV1 at all post-dose timepoints
To complete the evaluation of FEV1 and the potential for bronchoconstriction of the study treatment (number and percentage of subjects with a relative decrease from pre-dose in FEV1) | Day 1, Day 7, Week 4, Week 12
  Calculation of number and percentage of subjects with a relative decrease from pre-dose in FEV1 at each post-dose timpoint and at any post -dose timepoint > 15%
To complete the evaluation of FEV1 and the potential for bronchoconstriction of the study treatment (Absolute and relative changes from baseline in pre-dose FEV1) | Day 1, Day 7, Week 4, Week 12
  Absolute and relative changes from baseline in pre-dose FEV1 at all clinical visits
To complete the evaluation of FEV1 and the potential for bronchoconstriction of the study treatment (Change from pre-dose in FEV1) | Day 1, Day 7, Week 12
  Change from pre-dose in FEV1 AUC 0-2h
Peak expiratory flow (PEF) change from baseline at each inter-visit period over the entire treatment period | Inter-visit, over the entire 12 weeks treatment period
  Change from baseline at each inter-visit period and over the entire treatment period in morning and evening PEF
Percentage of days without intake of rescue medication. | Inter-visit, over the entire 12 weeks treatment period
  Change from baseline at each inter-visit period and over the entire treatment period in the percentage of days without intake of rescue medications
Change in the average daily use of rescue medication. | Inter-visit, over the entire 12 weeks treatment period
  Change from baseline at each inter-visit period and over the entire treatment period in the average daily use of rescue medication (number of inhalations/day)
Change on the average daily asthma symptoms. | Inter-visit, over the entire 12 weeks treatment period
  Change from baseline at each inter-visit period and over the entire treatment period in the average daily symptoms. Patients are asked to complete daily a questionnaire to collect this information and allow their asthma symptoms to be monitored.
Change from baseline in Asthma Control Questionnaire 7 (ACQ 7) score. | At each planned on site study visit, during the entire 12 weeks treatment period.
  ACQ 7 is a one week recall questionnaire including 6 questions to be completed by patients on a 7-points scale (0=no impairment, 6= maximum impairment) and 7th point capturing the FEV1 % predicted value (also scoring on a 7-point scale). Questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).

OTHER OUTCOMES:
To measure the safety and tolerability of CHF5993 pMDI HFA-152a in terms of Adverse Events (AEs) / Adverse Drug Reactions (ADRs). | Through study completion, an average of 1 year
  Number and percentage of subjects experiencing AEs, number and percentage of subjects experiencing at least one ADR and number and percentage of subjects experiencing at least one Treatment Emergent Adverse Events (TEAEs)
To measure the safety and tolerability of CHF5993 pMDI HFA-152a in terms of number of Adverse Events (AEs) of particular interest. | Through study completion, an average of 1 year
  Number of AEs for each of the following event: cough, dysphonia, paradoxical bronchospasm, hypersensitivity reactions, severe asthma Exacerbations
To measure the safety and tolerability of CHF5993 pMDI HFA-152a in terms of incident rate of Adverse Events (AEs) of particular interest. | Through study completion, an average of 1 year
  Incident rate for each of the following AE of particular interest: cough, dysphonia, paradoxical bronchospasm, hypersensitivity reactions, severe asthma Exacerbations.
To measure the safety and tolerability of CHF5993 pMDI HFA-152a in terms of rate ration of Adverse Events (AEs) of particular interest. | Through study completion, an average of 1 year
  Rate ratio between treatments for each of the following AE of particular interest: cough, dysphonia, paradoxical bronchospasm, hypersensitivity reactions, severe asthma Exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit, Langley Building, Wythenshawe Hospital
Locations (117):
- Bulgaria (18):
  - "IPSMCPP-D-R Veleva" EOOD, Burgas
  - Medical Center "Zdrave -1", Kozloduy
  - "AIPSMP Yuskyan Aliosman" Ltd, Momchilgrad
  - Ambulatory for Specialized Outpatient Medical Care - Individual Practice, Rousse
  - Specialized Hospital For Active Treatment Of Pneumo-Phthisiatric Diseases Dr. Dimitar Gramatikov - Ruse Ltd., Rousse
  - Specialized Hospital For Active Treatment Of Pneumo-Phthisiatric Diseases Dr. Dimitar Gramatikov, Rousse
  - Multiprofile Hospital For Active Treatment - Shumen AD,, Shumen
  - Diagnostic Consultative Centre 1-, Sliven
  - MHAT Sliven to MMA Sofia, Sliven
  - University First Multiprofile Hospital for Active Treatment -Sofia "St. Joan Krastilel" EAD, Sofia
  - Multiprofile Hospital For Active Treatment "Knyaginya Klementina" Sofia EAD,, Sofia
  - Medical Center Hera EOOD, 20 Klisura str., fl. 2,, Sofia
  - Multi-profile Hospital for Active Treatment Zdraveto 2012 Ltd.,, Sofia
  - Diagnostics and Consultation Center Convex EOOD, Sofia
  - "Medical Center Sun i Zdrave", Sofia
  - Medical Center "Syrtuin" Ltd, Sofia
  - Medical Center "New Rehabilitation Center" Ltd, Stara Zagora
  - ASMP MC Kissiovi Ltd., Varna
- Czechia (7):
  - Hornmed, s.r.o, Brno
  - Nemocnice Jihlava, Plicní oddělení, Jihlava
  - MediTrial s.r.o., Jindřichův Hradec
  - Pneumology dpt., Poliklinika Budějovická, MEDICON a.s., Prague
  - Pneumology dpt., Fakultní Thomayerova nemocnice, Prague
  - Prvni plicni ambulance s.r.o, Prague
  - Plicní středisko Teplice s.r.o., Teplice
- Georgia (9):
  - Geo Hospitals Gardabani Multiprofile Medical Centre, Gardabani
  - Geo Hospitals Gurjaani Multiprofile Medical Centre, Gurjaani
  - Geo Hospitals Sagarejo Multiprofile Medical Centre, Sagarejo
  - Medihelp Ltd, Samtredia
  - Imermedi-Imereti Regional Medical Center. (Terjolamedi) Ltd., T'erjola
  - Curatio, Jsc, Tbilisi
  - Geo Hospitals Tbilisi Multiprofile Medical Center, Tbilisi
  - First Medical Center LLC, Tbilisi
  - GEO HOSPITALS Zestaphoni Ambulatory Centre, Zestaponi
- Germany (16):
  - Studienpraxis Berlin-Brandenburg Cornelia Seelbinder Und Lennart Schaper GbR, Berlin
  - Lungenpraxis Hohenzollerndamm, Berlin
  - Klinische Forschung Berlin, Berlin
  - Policum Berlin Studien GmbH Friedenau, Berlin
  - Institut für Allergie- und Asthmaforschung, Berlin
  - Dr. med. Thomas Ginko Facharzt für Lungen- und Bronchialheilkunde, Bonn
  - Neudorfer Lungenpraxis, Duisburg
  - IKF Pneumologie Frankfurt Clinical Research Centre Respiratory Medicine IFS - Interdisziplinäres Facharztzentrum, Frankfurt
  - Athanasios Xanthopoulos Praxis für Pneumologie, Fürstenwalde
  - Praxis für Pneumologie und Allergologie, Leipzig
  - POIS Sachsen GmbH, Leipzig
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck
  - SMO Zentrum für klinische Studien, Magdeburg
  - Pneumologisches Studienzentrum München, München
  - Siteworks Prüfzentrum Schleswig GmbH, Schleswig
  - Lungenpraxis Witten, Witten
- "George Papanikolaou" General Hospital of Thessaloniki, Thessaloniki, Greece
- Hungary (6):
  - University of Debrecen, Infectology Clinic Pulmonary unit, Debrecen
  - Erzsébet Gondozóház, Gödöllő
  - BKS Research Kft.,, Hatvan
  - Revamed Kft, Nyíregyháza
  - INFER-MED Kft, Pécs
  - Árkádia Egészségközpont, Szombathely
- Italy (3):
  - Clinica Malattie Respiratorie e allergologia IRCCS Ospedale Policlinico San Martino, Genova
  - University of Messina, Allergy and Clinical Immunology Unit, Department of Experimental and Clinical Medicine, Messina
  - Azienda Ospedaliera dei colli - Ospedale Monaldi, Napoli
- Netherlands (3):
  - EB FlevoResearch BV, Almere Stad
  - Amphia Hospital, Breda
  - Gelre Hospitals Zutphen (Gelre ziekenhuizen Zutphen), Zutphen
- Poland (22):
  - Prywatny gabinet internistyczno-alergologiczny prof. Zenon Siergiejko, Bialystok
  - Centrum Medycyny Oddechowej, Mróz Spółka Jawna, Bialystok
  - Uniwersytet Medyczny w Bialymstoku Wydzial Nauk o Zdrowiu Klinika Alergologii i Chorób Wewnetrznych, Bialystok
  - Prywatna praktyka lekarska. Gabinet pediatryczno - alergologiczny, Bialystok
  - Vitamed Galaj I Cichomski Sp. J., Bydgoszcz
  - Centrum Nowoczesnych Terapii "Dobry Lekarz", Krakow
  - Private Health Care MEDYK-KRAK Sp. o.o., Krakow
  - Diamond Clinic Spółka z ograniczoną odpowiedzialnością, Krakow
  - Małopolskie Centrum Alergologii sp. z o.o., Krakow
  - ATOPIA Niepubliczny Zakład Opieki Zdrowotnej, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego, Lodz
  - Makowskie Centrum Medyczne MCM "Hamernia" Maków Podhalański, Maków Podhalański
  - Ostrowieckie Centrum Medyczne Spółka Cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Prywatny Gabinet Lekarski Małgorzata Pawlukiewicz, Rzeszów
  - Clinmedica Research Sp. Z O.O., Skierniewice
  - PULMAG Grzegorz Gąsior, Marzena Kociołek spółka cywilna, Sosnowiec
  - Centrum Medyczne Lucyna i Andrzej DymeK, Strzelce Opolskie
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z o. o., Tarnów
  - CLINICAL BEST SOLUTIONS Fiutkowski Sp. z o.o., Warsaw
  - Centrum Badań Klinicznych, Wroclaw
  - Michał Bogacki Dobrostan, Wroclaw
  - Lekarze Specjaliści - J. Małolepszy I Partnerzy, Wroclaw
- Romania (10):
  - Angisan Grup Srl, Bragadiru
  - Centrul Medical Sana (SANA S.R.L.), Bucharest
  - National Institute of Pneumology Marius Nasta, Bucharest
  - Medsana Bucharest Medical Center Srl, Bucharest
  - Spitalul Clinic de Pneumoftiziologie Leon Daniello, Cluj-Napoca
  - Spitalul clinic de Pneumoftiziologie Palazu Mare Constanta, Constanța
  - Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie "Victor Babeș" Craiova, Craiova
  - Spital Judetean de Urgenta Bihor, Oradea
  - Clinical Hospital of Infectious Diseases and Pneumophysiology Dr.Victor Babeș Timișoara, Timișoara
  - Clinical Hospital of Infectious Diseases and Pneumophysiology, Timișoara
- Serbia (7):
  - Clinic for Pulmonary Diseases, University Clinical center of Serbia, Belgrade
  - Municipal Institute for lung diseases and tuberculosis, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina., Kamenica
  - Clinic for Pulmonology, University Clinical Center Kragujevac., Kragujevac
  - Clinic for Pulmonology, University Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Niš Clinic for Lung Diseases, Niš
  - Užice General Hospital Miloša Obrenovića 17., Užice
- Slovakia (6):
  - Poliklinika ČK PLUS Alian s.r.o, Bardejov
  - Pľucna ambulancia MUDr. Miroslava Undesser, Dunajská Streda
  - Nemocnica s poliklinikou Š. Kukuru Michalovce, Michalovce
  - Pľúcna ambulacia - MUDr. Slavomír Hrebenár, Spišská Nová Ves
  - IMUNOALERGOLÓGIA JZ, s.r.o., Žilina
  - KOMA Kardioprax, s.r.o., Žilina
- Spain (4):
  - Hospital General Universitario de Castellón, Castellon
  - Giromed Institute Parc Científic i Tecnològic Universitat de Girona, Girona
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario Universitario de Santiago Hospital Clínico Universitario de Santiago, Santiago de Compostela
- United Kingdom (5):
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Queen Mary University of London, London
  - Guy's & St Thomas'NHS Foundation Trust of Royal Brompton Hospital, London
  - Medicines Evaluation Unit, Langley Building, Wythenshawe Hospital, Manchester
  - Portsmouth Hospitals University NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No